CLINICAL TRIAL: NCT00145457
Title: A Multicentre Study on the Capacity of the IGF-1 Stimulation Test to Predict the Growth Promoting Effect of Standard and High Doses of Genotonorm® in Prepubertal Children With Growth Hormone Deficiency.
Brief Title: IGF1 Generation Test
Acronym: CAREL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 307-MET-9002-040; A6281023
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 2007-05

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Blood Specimen Collection; X-Rays

INTERVENTIONS:
Procedure: Blood sample
Procedure: Radiography

SUMMARY:
To assess the predictive value of the short term IGF-1 stimulation test, based on IGF-1 changes, on the 24 months growth response to 2 different doses of GH in patients with conventional GH deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged of more than 4 years.
* GHD defined as a peak GH level < 20 mUI/ml at two different pharmacological GH provocative tests including one done with two pharmacological agents and both performed within the year before the inclusion, according to the current recommendations of the French Health Authorities

Exclusion Criteria:

* Previous treatment with GH
* Ongoing pharmacological treatment with steroids except if corresponding to substitutive therapy

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82
Dates: Start 2001-04; Study Completion 2005-01

PRIMARY OUTCOMES:
Change of height standard deviation score after 24 months of treatment according to the short term response of plasma IGF1 to Genotonorm.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- France (8):
  - Pfizer Investigational Site, BesanÃ§on
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Dunkirk
  - Pfizer Investigational Site, Limoges
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Tarbes
  - Pfizer Investigational Site, Toulouse